CLINICAL TRIAL: NCT04615910
Title: A GLP-1 Receptor PET Imaging Substudy Within the VER-A-T1D Trial Investigating the Effects on Beta Cell Mass
Acronym: Ver-A-image
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Medical University of Vienna (Other); Bart's London (Unknown); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20201013
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
Keywords: Verapamil; Type 1 Diabetes Mellitus; exendin; Beta cell mass; PET imaging
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Type 1 Diabetes Mellitus
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verapamil (Experimental): Patients treated with Verapamil within the Ver-A-T1D trial
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT
- Placebo (Placebo Comparator): Patients treated with placebo within the Ver-A-T1D trial
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT

INTERVENTIONS:
Radiation: 68Ga-NODAGA-exendin-4 PET/CT — 68Ga-NODAGA-exendin-4 PET/CT

SUMMARY:
The goal of the trial is to measure pancreatic uptake of 68Ga-NODAGA-exendin by PET/CT for detection of intra-individual differences in beta cell mass before and after treatment with Verapamil.

DETAILED DESCRIPTION:
The VER-A-T1D (Verapamil SR in adults with Type 1 Diabetes) study is an intervention study within the INNODIA project (an Innovative Medicines Initiative consortium (IMI-2), established through Horizon 2020 initiative of the European Union, involving academic, industry and charitable partners).

In the VER-A-T1D study, the effects of treatment of newly diagnosed patients with T1D with Verapamil will be evaluated. Verapamil appears to protect beta cell function, an effect that could in part be caused by protection against beta cell apoptosis. GLP-1 receptors are expressed in high densities in beta cells. Exendin, a GLP-1 receptor agonist, can be labeled with radionuclides and thus be utilized for visualization of beta cells in vivo by positron emission tomography (PET). This technology has been demonstrated to deliver quantitative information of the radiotracer uptake in the pancreas demonstrating a linear correlation with beta cell mass. In VER-A-T1D, we propose to measure beta cell mass at the time points of inclusion and at evaluation after 12 months. If verapamil protects beta cells against apoptosis, we expect that the uptake of the radiotracer will be higher at 12 months in comparison to the first measurement in the treatment group. The study will be a substudy to VER-A-T1D.

ELIGIBILITY:
Inclusion Criteria:

* • Have given written informed consent
* • Age ≥18 and <45 at consent
* • Must have a diagnosis of T1D of within 6 weeks duration at screening (date of the first insulin
* injection)
* • Must have at least one or more diabetes-related autoantibodies present at screening
* • Must have random C-peptide levels ≥200 pmol/L measured at screening
* • Be willing to comply with intensive diabetes management

Exclusion Criteria:

* Treatment with synthetic Exendin (Exenatide, Byetta®) or Dipeptidyl-Peptidase IV inhibitors (to exclude interferences with imaging, specifically mentioned although in principle part of exclusion criteria of VER-A-T1D)
* Renal disease defined as MDRD <40 ml/min/1.73 m2
* Pregnancy or the wish to become pregnant within 2 months after the second PET/CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic 68Ga-exendin uptake | Change from time of inclusion to 12 months into treatment
  the total pancreatic uptake of 68Ga-NODAGA-exendin by PET/CT for determination of beta cell mass

SECONDARY OUTCOMES:
Correlation of 68Ga-exendin uptake and C-peptide | 12 months into treatment
  • Changes in 68Ga-NODAGA-exendin pancreas uptake in realtion to changes in C-peptide measurements.
relative 68Ga-exendin uptake | 12 months into treatment
  • Differences in 68Ga-NODAGA-exendin uptake between individuals and between the two timepoints of imaging intra-individually

CONTACTS AND LOCATIONS:
Locations (2):
- University of Vienna, Vienna, Austria
- Assistance Publique hopitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No